CLINICAL TRIAL: NCT00000125
Title: Ocular Hypertension Treatment Study (OHTS)
Acronym: OHTS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NEI-24; 5U10EY009307-16 (NIH); 5U10EY009341-14 (NIH)
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Results first posted 2015-03-19 (Estimated); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Ocular Hypertension; Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Observation (No Intervention): Close Observation.
- Treatment (Other): Participants treated with commercially available topical ocular hypotensive eye drops.
  Interventions: Drug: Topical ocular hypotensive eye drops.

INTERVENTIONS:
Drug: Topical ocular hypotensive eye drops. — Topical ocular hypotensive eye drops.
  Arms: Treatment

SUMMARY:
To determine whether medical reduction of intraocular pressure prevents or delays the onset of glaucomatous visual field loss and/or optic disc damage in ocular hypertensive participants judged to be at moderate risk for developing open-angle glaucoma.

To produce natural history data to assist in identifying patients at most risk for developing open-angle glaucoma and those most likely to benefit from early medical treatment.

To quantify risk factors for developing open-angle glaucoma among ocular hypertensive individuals.

DETAILED DESCRIPTION:
OHTS Phase 3 will re-examine study participants 20 plus years after enrollment to document clinical status and the incidence and severity of self-reported functional limitations. The 279 participants who developed POAG in OHTS Phase 1 or 2 will have more than 10 years of post-POAG follow-up by Phase 3. The timing of re-examination at 20 years is meaningful because 20 years approaches the median life expectancy of OHT patients in their 60's and 70's and half the median life expectancy of patients in their 40's and 50's. For the first time, patients with ocular hypertension and clinicians will have high quality data about the long-term risk of developing POAG and functional limitations associated with the disease. These data will facilitate patient-centered care so that patients and clinicians can decide on the appropriate frequency of tests and examinations and the potential benefit of preventative treatment.

Glaucoma is one of the leading causes of blindness in the United States and other industrialized countries. It is estimated that 2 million people in the United States have glaucoma and that 80,000 of these individuals are legally blind from the disease. Among African Americans, glaucoma is now recognized as the leading cause of blindness.

Elevated intraocular pressure (IOP), a common condition affecting 3 to 6 million people in the United States, is thought to be the leading risk factor for development of open-angle glaucoma. There is no consensus that medical reduction of intraocular pressure prevents or delays the onset of visual field and/or optic nerve damage in ocular hypertensive subjects.

Despite the lack of convincing evidence for the efficacy of medical treatment in ocular hypertension, approximately 1.5 million glaucoma suspects in the United States are being treated with costly ocular hypotensive medications that carry the potential for serious and even life-threatening side effects.

Clearly, there is a need for a well-controlled clinical trial to determine whether medical reduction of IOP can prevent or delay the onset of glaucomatous damage in ocular hypertensive subjects. Only then can clinicians and patients make rational choices and health care planners ensure that limited medical resources are being allocated in a safe and cost-effective manner.

The Ocular Hypertension Treatment Study (OHTS) is a long-term, randomized, controlled multicenter clinical trial. Ocular hypertensive subjects judged to be at moderate risk of developing primary open-angle glaucoma are randomly assigned to either close observation only or a stepped medical regimen. Medical treatment consists of all commercially available topical ocular hypotensive eye drops.

After completion of baseline measures (IOP, visual fields, disc photos) and randomization, the subjects are followed for a minimum of 5 years with automated threshold central static perimetry (Humphrey program 30-2) twice yearly and stereoscopic optic disc photographs once yearly. Study end points are reproducible visual field loss and/or progressive optic disc damage in either eye of a patient attributed to glaucoma by a Masked Endpoint Committee. All visual fields and optic disc photographs are read in a masked fashion in Reading Centers.

In the 1991 Baltimore Eye Survey, African Americans were shown to have a prevalence of open-angle glaucoma four to five times higher than whites. Given this high prevalence of glaucoma in the African American population, it is important to recruit and follow an adequate sample of African American subjects in the trial (approximately 25 percent of the total patient sample).

At the conclusion of this study, practitioners should be able to make reasonable estimates of risk for individual ocular hypertensive patients and to determine which ocular hypertensive individuals are most likely to benefit from early prophylactic medical treatment.

ELIGIBILITY:
Men and nonpregnant women between the ages of 40 and 80 with IOP greater than or equal to 24 mm Hg but less than or equal to 32 mm Hg in at least one eye and IOP greater than or equal to 21 but less than or equal to 32 mm Hg in the fellow eye, as well as normal visual fields and optic discs are eligible for the trial. Patients presenting with best-corrected visual acuity worse than 20/40 in either eye, previous intraocular surgery, a life-threatening or debilitating disease, secondary causes of elevated IOP, angle-closure glaucoma or anatomically narrow angles, other diseases that can cause visual field loss, background diabetic retinopathy, optic disc abnormalities that can produce visual field loss or obscure the interpretation of the optic disc, or unwillingness to undergo random assignment are excluded from the trial.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1636 (Actual)
Dates: Start 1994-02 (Actual); Primary Completion 2002-06 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Kass, MD, Study Chair — Washington University Department of Ophthalmology and Visual Sciences

REFERENCES:
- [Background] Gordon MO, Kass MA. The Ocular Hypertension Treatment Study: design and baseline description of the participants. Arch Ophthalmol. 1999 May;117(5):573-83. doi: 10.1001/archopht.117.5.573. PMID 10326953
- [Background] Keltner JL, Johnson CA, Quigg JM, Cello KE, Kass MA, Gordon MO. Confirmation of visual field abnormalities in the Ocular Hypertension Treatment Study. Ocular Hypertension Treatment Study Group. Arch Ophthalmol. 2000 Sep;118(9):1187-94. doi: 10.1001/archopht.118.9.1187. PMID 10980763
- [Background] Piltz J, Gross R, Shin DH, Beiser JA, Dorr DA, Kass MA, Gordon MO. Contralateral effect of topical beta-adrenergic antagonists in initial one-eyed trials in the ocular hypertension treatment study. Am J Ophthalmol. 2000 Oct;130(4):441-53. doi: 10.1016/s0002-9394(00)00527-4. PMID 11024416
- [Background] Brandt JD, Beiser JA, Kass MA, Gordon MO. Central corneal thickness in the Ocular Hypertension Treatment Study (OHTS). Ophthalmology. 2001 Oct;108(10):1779-88. doi: 10.1016/s0161-6420(01)00760-6. PMID 11581049
- [Background] Feuer WJ, Parrish RK 2nd, Schiffman JC, Anderson DR, Budenz DL, Wells MC, Hess DJ, Kass MA, Gordon MO. The Ocular Hypertension Treatment Study: reproducibility of cup/disk ratio measurements over time at an optic disc reading center. Am J Ophthalmol. 2002 Jan;133(1):19-28. doi: 10.1016/s0002-9394(01)01338-1. PMID 11755836
- [Background] Johnson CA, Keltner JL, Cello KE, Edwards M, Kass MA, Gordon MO, Budenz DL, Gaasterland DE, Werner E; Ocular Hypertension Study Group. Baseline visual field characteristics in the ocular hypertension treatment study. Ophthalmology. 2002 Mar;109(3):432-7. doi: 10.1016/s0161-6420(01)00948-4. PMID 11874743
- [Background] Kass MA, Heuer DK, Higginbotham EJ, Johnson CA, Keltner JL, Miller JP, Parrish RK 2nd, Wilson MR, Gordon MO. The Ocular Hypertension Treatment Study: a randomized trial determines that topical ocular hypotensive medication delays or prevents the onset of primary open-angle glaucoma. Arch Ophthalmol. 2002 Jun;120(6):701-13; discussion 829-30. doi: 10.1001/archopht.120.6.701. PMID 12049574
- [Background] Gordon MO, Beiser JA, Brandt JD, Heuer DK, Higginbotham EJ, Johnson CA, Keltner JL, Miller JP, Parrish RK 2nd, Wilson MR, Kass MA. The Ocular Hypertension Treatment Study: baseline factors that predict the onset of primary open-angle glaucoma. Arch Ophthalmol. 2002 Jun;120(6):714-20; discussion 829-30. doi: 10.1001/archopht.120.6.714. PMID 12049575
- [Background] Keltner JL, Johnson CA, Cello KE, Edwards MA, Bandermann SE, Kass MA, Gordon MO; Ocular Hypertension Treatment Study Group. Classification of visual field abnormalities in the ocular hypertension treatment study. Arch Ophthalmol. 2003 May;121(5):643-50. doi: 10.1001/archopht.121.5.643. PMID 12742841
- [Background] Zangwill LM, Weinreb RN, Berry CC, Smith AR, Dirkes KA, Coleman AL, Piltz-Seymour JR, Liebmann JM, Cioffi GA, Trick G, Brandt JD, Gordon MO, Kass MA; Confocal Scanning Laser Ophthalmoscopy Ancillary Study to the Ocular Hypertension Treatment Study. Racial differences in optic disc topography: baseline results from the confocal scanning laser ophthalmoscopy ancillary study to the ocular hypertension treatment study. Arch Ophthalmol. 2004 Jan;122(1):22-8. doi: 10.1001/archopht.122.1.22. PMID 14718290
- [Background] Zangwill LM, Weinreb RN, Berry CC, Smith AR, Dirkes KA, Liebmann JM, Brandt JD, Trick G, Cioffi GA, Coleman AL, Piltz-Seymour JR, Gordon MO, Kass MA; OHTS CSLO Ancillary Study Group. The confocal scanning laser ophthalmoscopy ancillary study to the ocular hypertension treatment study: study design and baseline factors. Am J Ophthalmol. 2004 Feb;137(2):219-27. doi: 10.1016/j.ajo.2003.08.031. PMID 14962409
- [Background] Higginbotham EJ, Gordon MO, Beiser JA, Drake MV, Bennett GR, Wilson MR, Kass MA; Ocular Hypertension Treatment Study Group. The Ocular Hypertension Treatment Study: topical medication delays or prevents primary open-angle glaucoma in African American individuals. Arch Ophthalmol. 2004 Jun;122(6):813-20. doi: 10.1001/archopht.122.6.813. PMID 15197055
- [Background] Coleman AL, Gordon MO, Beiser JA, Kass MA; Ocular Hypertension Treatment Study. Baseline risk factors for the development of primary open-angle glaucoma in the Ocular Hypertension Treatment Study. Am J Ophthalmol. 2004 Oct;138(4):684-5. doi: 10.1016/j.ajo.2004.05.030. PMID 15488816
- [Background] Brandt JD, Beiser JA, Gordon MO, Kass MA; Ocular Hypertension Treatment Study (OHTS) Group. Central corneal thickness and measured IOP response to topical ocular hypotensive medication in the Ocular Hypertension Treatment Study. Am J Ophthalmol. 2004 Nov;138(5):717-22. doi: 10.1016/j.ajo.2004.07.036. PMID 15531304
- [Background] Kass MA, Gordon MO, Kymes SM. Incorporating the results of the Ocular Hypertension Treatment Study into clinical practice. Arch Ophthalmol. 2005 Jul;123(7):1021-2. doi: 10.1001/archopht.123.7.1021-b. No abstract available. PMID 16009857
- [Background] Zangwill LM, Weinreb RN, Beiser JA, Berry CC, Cioffi GA, Coleman AL, Trick G, Liebmann JM, Brandt JD, Piltz-Seymour JR, Dirkes KA, Vega S, Kass MA, Gordon MO. Baseline topographic optic disc measurements are associated with the development of primary open-angle glaucoma: the Confocal Scanning Laser Ophthalmoscopy Ancillary Study to the Ocular Hypertension Treatment Study. Arch Ophthalmol. 2005 Sep;123(9):1188-97. doi: 10.1001/archopht.123.9.1188. PMID 16157798
- [Background] Keltner JL, Johnson CA, Levine RA, Fan J, Cello KE, Kass MA, Gordon MO. Normal visual field test results following glaucomatous visual field end points in the Ocular Hypertension Treatment Study. Arch Ophthalmol. 2005 Sep;123(9):1201-6. doi: 10.1001/archopht.123.9.1201. PMID 16157799
- [Background] Parrish RK 2nd, Schiffman JC, Feuer WJ, Anderson DR, Budenz DL, Wells-Albornoz MC, Vandenbroucke R, Kass MA, Gordon MO; Ocular Hypertension Treatment Study Group. Test-retest reproducibility of optic disk deterioration detected from stereophotographs by masked graders. Am J Ophthalmol. 2005 Oct;140(4):762-4. doi: 10.1016/j.ajo.2005.04.044. PMID 16226544
- [Background] Kymes SM, Kass MA, Anderson DR, Miller JP, Gordon MO; Ocular Hypertension Treatment Study Group (OHTS). Management of ocular hypertension: a cost-effectiveness approach from the Ocular Hypertension Treatment Study. Am J Ophthalmol. 2006 Jun;141(6):997-1008. doi: 10.1016/j.ajo.2006.01.019. PMID 16765666
- [Background] Levine RA, Demirel S, Fan J, Keltner JL, Johnson CA, Kass MA; Ocular Hypertension Treatment Study Group. Asymmetries and visual field summaries as predictors of glaucoma in the ocular hypertension treatment study. Invest Ophthalmol Vis Sci. 2006 Sep;47(9):3896-903. doi: 10.1167/iovs.05-0469. PMID 16936102
- [Background] Keltner JL, Johnson CA, Anderson DR, Levine RA, Fan J, Cello KE, Quigley HA, Budenz DL, Parrish RK, Kass MA, Gordon MO; Ocular Hypertension Treatment Study Group. The association between glaucomatous visual fields and optic nerve head features in the Ocular Hypertension Treatment Study. Ophthalmology. 2006 Sep;113(9):1603-12. doi: 10.1016/j.ophtha.2006.05.061. PMID 16949445
- [Background] Herman DC, Gordon MO, Beiser JA, Chylack LT Jr, Lamping KA, Schein OD, Soltau JB, Kass MA; Ocular Hypertension Treatment Study (OHTS) Group. Topical ocular hypotensive medication and lens opacification: evidence from the ocular hypertension treatment study. Am J Ophthalmol. 2006 Nov;142(5):800-10. doi: 10.1016/j.ajo.2006.06.052. PMID 17056362
- [Background] Budenz DL, Anderson DR, Feuer WJ, Beiser JA, Schiffman J, Parrish RK 2nd, Piltz-Seymour JR, Gordon MO, Kass MA; Ocular Hypertension Treatment Study Group. Detection and prognostic significance of optic disc hemorrhages during the Ocular Hypertension Treatment Study. Ophthalmology. 2006 Dec;113(12):2137-43. doi: 10.1016/j.ophtha.2006.06.022. Epub 2006 Sep 25. PMID 16996592
- [Background] Ocular Hypertension Treatment Study Group; European Glaucoma Prevention Study Group; Gordon MO, Torri V, Miglior S, Beiser JA, Floriani I, Miller JP, Gao F, Adamsons I, Poli D, D'Agostino RB, Kass MA. Validated prediction model for the development of primary open-angle glaucoma in individuals with ocular hypertension. Ophthalmology. 2007 Jan;114(1):10-9. doi: 10.1016/j.ophtha.2006.08.031. Epub 2006 Nov 7. PMID 17095090
- [Background] Mansberger SL, Hughes BA, Gordon MO, Spaner SD, Beiser JA, Cioffi GA, Kass MA; Ocular Hypertension Treatment Study Group. Comparison of initial intraocular pressure response with topical beta-adrenergic antagonists and prostaglandin analogues in African American and white individuals in the Ocular Hypertension Treatment Study. Arch Ophthalmol. 2007 Apr;125(4):454-9. doi: 10.1001/archopht.125.4.454. PMID 17420364
- [Background] Keltner JL, Johnson CA, Cello KE, Bandermann SE, Fan J, Levine RA, Kass MA, Gordon MO; Ocular Hypertension Treatment Study Group. Visual field quality control in the Ocular Hypertension Treatment Study (OHTS). J Glaucoma. 2007 Dec;16(8):665-9. doi: 10.1097/IJG.0b013e318057526d. PMID 18091452
- [Background] Gordon MO, Beiser JA, Kass MA; Ocular Hypertension Treatment Study Group. Is a history of diabetes mellitus protective against developing primary open-angle glaucoma? Arch Ophthalmol. 2008 Feb;126(2):280-1. doi: 10.1001/archophthalmol.2007.35. No abstract available. PMID 18268230
- [Background] Kass MA, Gordon MO; Ocular Hypertension Treatment Study Group. Diabetes and glaucoma. Arch Ophthalmol. 2008 May;126(5):746-7. doi: 10.1001/archopht.126.5.746-b. No abstract available. PMID 18474807
- [Background] Brandt JD, Gordon MO, Beiser JA, Lin SC, Alexander MY, Kass MA; Ocular Hypertension Treatment Study Group. Changes in central corneal thickness over time: the ocular hypertension treatment study. Ophthalmology. 2008 Sep;115(9):1550-6, 1556.e1. doi: 10.1016/j.ophtha.2008.02.001. Epub 2008 Apr 18. PMID 18378313
- [Background] Ocular Hypertension Treatment Study Group and the European Glaucoma Prevention Study Group. The accuracy and clinical application of predictive models for primary open-angle glaucoma in ocular hypertensive individuals. Ophthalmology. 2008 Nov;115(11):2030-6. doi: 10.1016/j.ophtha.2008.06.036. Epub 2008 Sep 18. PMID 18801578
- [Background] Bhorade AM, Gordon MO, Wilson B, Weinreb RN, Kass MA; Ocular Hypertension Treatment Study Group. Variability of intraocular pressure measurements in observation participants in the ocular hypertension treatment study. Ophthalmology. 2009 Apr;116(4):717-24. doi: 10.1016/j.ophtha.2008.12.036. Epub 2009 Feb 25. PMID 19243824
- [Background] Barnett EM, Fantin A, Wilson BS, Kass MA, Gordon MO; Ocular Hypertension Treatment Study Group. The incidence of retinal vein occlusion in the ocular hypertension treatment study. Ophthalmology. 2010 Mar;117(3):484-8. doi: 10.1016/j.ophtha.2009.08.022. Epub 2010 Jan 19. PMID 20031222
- [Background] Kymes SM, Plotzke MR, Kass MA, Boland MV, Gordon MO. Effect of patient's life expectancy on the cost-effectiveness of treatment for ocular hypertension. Arch Ophthalmol. 2010 May;128(5):613-8. doi: 10.1001/archophthalmol.2010.83. PMID 20457984
- [Background] Weinreb RN, Zangwill LM, Jain S, Becerra LM, Dirkes K, Piltz-Seymour JR, Cioffi GA, Trick GL, Coleman AL, Brandt JD, Liebmann JM, Gordon MO, Kass MA; OHTS CSLO Ancillary Study Group. Predicting the onset of glaucoma: the confocal scanning laser ophthalmoscopy ancillary study to theOcular Hypertension Treatment Study. Ophthalmology. 2010 Sep;117(9):1674-83. doi: 10.1016/j.ophtha.2010.03.044. Epub 2010 Jul 14. PMID 20633931
- [Background] Bhorade AM, Wilson BS, Gordon MO, Palmberg P, Weinreb RN, Miller E, Chang RT, Kass MA; Ocular Hypertension Treatment Study Group. The utility of the monocular trial: data from the ocular hypertension treatment study. Ophthalmology. 2010 Nov;117(11):2047-54. doi: 10.1016/j.ophtha.2010.02.020. Epub 2010 Aug 12. PMID 20619460
- [Background] Artes PH, Chauhan BC, Keltner JL, Cello KE, Johnson CA, Anderson DR, Gordon MO, Kass MA; Ocular Hypertension Treatment Study Group. Longitudinal and cross-sectional analyses of visual field progression in participants of the Ocular Hypertension Treatment Study. Arch Ophthalmol. 2010 Dec;128(12):1528-32. doi: 10.1001/archophthalmol.2010.292. PMID 21149774
- [Background] Gao F, Miller JP, Xiong C, Beiser JA, Gordon M; The Ocular Hypertension Treatment Study (OHTS) Group. A joint-modeling approach to assess the impact of biomarker variability on the risk of developing clinical outcome. Stat Methods Appt. 2011 Mar 1;20(1):83-100. doi: 10.1007/s10260-010-0150-z. PMID 21339862
- [Background] Gao F, Miller JP, Miglior S, Beiser JA, Torri V, Kass MA, Gordon MO. A Joint Model for Prognostic Effect of Biomarker Variability on Outcomes: long-term intraocular pressure (IOP) fluctuation on the risk of developing primary open-angle glaucoma (POAG). JP J Biostat. 2011 May 1;5(2):73-96. PMID 22180704
- [Background] Gordon MO, Gao F, Beiser JA, Miller JP, Kass MA. The 10-year incidence of glaucoma among patients with treated and untreated ocular hypertension. Arch Ophthalmol. 2011 Dec;129(12):1630-1. doi: 10.1001/archophthalmol.2011.337. No abstract available. PMID 22159688
- [Background] Demirel S, De Moraes CG, Gardiner SK, Liebmann JM, Cioffi GA, Ritch R, Gordon MO, Kass MA; Ocular Hypertension Treatment Study Group. The rate of visual field change in the ocular hypertension treatment study. Invest Ophthalmol Vis Sci. 2012 Jan 25;53(1):224-7. doi: 10.1167/iovs.10-7117. PMID 22159015
- [Background] Brandt JD, Gordon MO, Gao F, Beiser JA, Miller JP, Kass MA; Ocular Hypertension Treatment Study Group. Adjusting intraocular pressure for central corneal thickness does not improve prediction models for primary open-angle glaucoma. Ophthalmology. 2012 Mar;119(3):437-42. doi: 10.1016/j.ophtha.2011.03.018. Epub 2011 Jun 25. PMID 21705084
- [Background] De Moraes CG, Demirel S, Gardiner SK, Liebmann JM, Cioffi GA, Ritch R, Gordon MO, Kass MA; Ocular Hypertension Treatment Study Group. Effect of treatment on the rate of visual field change in the ocular hypertension treatment study observation group. Invest Ophthalmol Vis Sci. 2012 Apr 2;53(4):1704-9. doi: 10.1167/iovs.11-8186. PMID 22395889
- [Background] Kymes SM, Lambert DL, Lee PP, Musch DC, Siegfried CJ, Kotak SV, Stwalley DL, Fain J, Johnson C, Gordon MO. The development of a decision analytic model of changes in mean deviation in people with glaucoma: the COA model. Ophthalmology. 2012 Jul;119(7):1367-74. doi: 10.1016/j.ophtha.2012.01.054. Epub 2012 Apr 25. PMID 22537616
- [Background] Mansberger SL, Gordon MO, Jampel H, Bhorade A, Brandt JD, Wilson B, Kass MA; Ocular Hypertension Treatment Study Group. Reduction in intraocular pressure after cataract extraction: the Ocular Hypertension Treatment Study. Ophthalmology. 2012 Sep;119(9):1826-31. doi: 10.1016/j.ophtha.2012.02.050. Epub 2012 May 16. PMID 22608478
- [Background] Gardiner SK, Demirel S, De Moraes CG, Liebmann JM, Cioffi GA, Ritch R, Gordon MO, Kass MA; Ocular Hypertension Treatment Study Group. Series length used during trend analysis affects sensitivity to changes in progression rate in the ocular hypertension treatment study. Invest Ophthalmol Vis Sci. 2013 Feb 15;54(2):1252-9. doi: 10.1167/iovs.12-10218. PMID 23349433
- [Background] Zangwill LM, Jain S, Dirkes K, He F, Medeiros FA, Trick GL, Brandt JD, Cioffi GA, Coleman AL, Liebmann JM, Piltz-Seymour JR, Gordon MO, Kass MA, Weinreb RN; Confocal Scanning Laser Ophthalmoscopy Ancillary Study to the Ocular Hypertension Treatment Study. The rate of structural change: the confocal scanning laser ophthalmoscopy ancillary study to the ocular hypertension treatment study. Am J Ophthalmol. 2013 Jun;155(6):971-82. doi: 10.1016/j.ajo.2013.01.020. Epub 2013 Mar 14. PMID 23497845
- [Background] Gardiner SK, Demirel S, Gordon MO, Kass MA; Ocular Hypertension Treatment Study Group. Seasonal changes in visual field sensitivity and intraocular pressure in the ocular hypertension treatment study. Ophthalmology. 2013 Apr;120(4):724-30. doi: 10.1016/j.ophtha.2012.09.056. Epub 2013 Jan 26. PMID 23357622
- [Background] De Moraes CG, Demirel S, Gardiner SK, Liebmann JM, Cioffi GA, Ritch R, Gordon MO, Kass MA. Rate of visual field progression in eyes with optic disc hemorrhages in the ocular hypertension treatment study. Arch Ophthalmol. 2012 Dec;130(12):1541-6. doi: 10.1001/jamaophthalmol.2013.1137. PMID 23229692
- [Background] Baratz KH, Nau CB, Winter EJ, McLaren JW, Hodge DO, Herman DC, Bourne WM. Effects of glaucoma medications on corneal endothelium, keratocytes, and subbasal nerves among participants in the ocular hypertension treatment study. Cornea. 2006 Oct;25(9):1046-52. doi: 10.1097/01.ico.0000230499.07273.c5. PMID 17133051
- [Background] Savatovsky E, Mwanza JC, Budenz DL, Feuer WJ, Vandenbroucke R, Schiffman JC, Anderson DR; Ocular Hypertension Treatment Study. Longitudinal changes in peripapillary atrophy in the ocular hypertension treatment study: a case-control assessment. Ophthalmology. 2015 Jan;122(1):79-86. doi: 10.1016/j.ophtha.2014.07.033. Epub 2014 Sep 7. PMID 25208858
- [Background] Christopher M, Abramoff MD, Tang L, Gordon MO, Kass MA, Budenz DL, Fingert JH, Scheetz TE. Stereo Photo Measured ONH Shape Predicts Development of POAG in Subjects With Ocular Hypertension. Invest Ophthalmol Vis Sci. 2015 Jul;56(8):4470-9. doi: 10.1167/iovs.14-16142. PMID 26193923
- [Background] Gao F, Miller JP, Beiser JA, Xiong C, Gordon MO. Predicting Clinical Binary Outcome Using Multivariate Longitudinal Data: Application to Patients with Newly Diagnosed Primary Open-Angle Glaucoma. J Biom Biostat. 2015 Oct;6(4):254. doi: 10.4172/2155-6180.1000254. Epub 2015 Oct 26. PMID 26904374
- [Background] Schaefer JL, Lukowski ZL, Meyer AM, Leoncavallo AJ, Greer A, Martorana GM, Zou B, Shuster JJ, Sherwood MB. Comparing Glaucomatous Disc Change Using Stereo Disc Viewing and the MatchedFlicker Software Program in Ophthalmologists-in-Training. Am J Ophthalmol. 2016 Jul;167:88-95. doi: 10.1016/j.ajo.2016.03.031. Epub 2016 Mar 31. PMID 27038890
- [Background] Scheetz TE, Faga B, Ortega L, Roos BR, Gordon MO, Kass MA, Wang K, Fingert JH. Glaucoma Risk Alleles in the Ocular Hypertension Treatment Study. Ophthalmology. 2016 Dec;123(12):2527-2536. doi: 10.1016/j.ophtha.2016.08.036. Epub 2016 Oct 1. PMID 27707548
- [Background] Khawaja AP, Cooke Bailey JN, Kang JH, Allingham RR, Hauser MA, Brilliant M, Budenz DL, Christen WG, Fingert J, Gaasterland D, Gaasterland T, Kraft P, Lee RK, Lichter PR, Liu Y, Medeiros F, Moroi SE, Richards JE, Realini T, Ritch R, Schuman JS, Scott WK, Singh K, Sit AJ, Vollrath D, Wollstein G, Zack DJ, Zhang K, Pericak-Vance M, Weinreb RN, Haines JL, Pasquale LR, Wiggs JL. Assessing the Association of Mitochondrial Genetic Variation With Primary Open-Angle Glaucoma Using Gene-Set Analyses. Invest Ophthalmol Vis Sci. 2016 Sep 1;57(11):5046-5052. doi: 10.1167/iovs.16-20017. PMID 27661856
- [Background] Bailey JN, Loomis SJ, Kang JH, Allingham RR, Gharahkhani P, Khor CC, Burdon KP, Aschard H, Chasman DI, Igo RP Jr, Hysi PG, Glastonbury CA, Ashley-Koch A, Brilliant M, Brown AA, Budenz DL, Buil A, Cheng CY, Choi H, Christen WG, Curhan G, De Vivo I, Fingert JH, Foster PJ, Fuchs C, Gaasterland D, Gaasterland T, Hewitt AW, Hu F, Hunter DJ, Khawaja AP, Lee RK, Li Z, Lichter PR, Mackey DA, McGuffin P, Mitchell P, Moroi SE, Perera SA, Pepper KW, Qi Q, Realini T, Richards JE, Ridker PM, Rimm E, Ritch R, Ritchie M, Schuman JS, Scott WK, Singh K, Sit AJ, Song YE, Tamimi RM, Topouzis F, Viswanathan AC, Verma SS, Vollrath D, Wang JJ, Weisschuh N, Wissinger B, Wollstein G, Wong TY, Yaspan BL, Zack DJ, Zhang K, Study EN; ANZRAG Consortium; Weinreb RN, Pericak-Vance MA, Small K, Hammond CJ, Aung T, Liu Y, Vithana EN, MacGregor S, Craig JE, Kraft P, Howell G, Hauser MA, Pasquale LR, Haines JL, Wiggs JL. Genome-wide association analysis identifies TXNRD2, ATXN2 and FOXC1 as susceptibility loci for primary open-angle glaucoma. Nat Genet. 2016 Feb;48(2):189-94. doi: 10.1038/ng.3482. Epub 2016 Jan 11. PMID 26752265
- [Background] Budenz DL, Huecker JB, Gedde SJ, Gordon M, Kass M; Ocular Hypertension Treatment Study Group. Thirteen-Year Follow-up of Optic Disc Hemorrhages in the Ocular Hypertension Treatment Study. Am J Ophthalmol. 2017 Feb;174:126-133. doi: 10.1016/j.ajo.2016.10.023. Epub 2016 Nov 7. PMID 27832941
- [Background] Schaefer JL, Meyer AM, Rodgers CD, Rosenberg NC, Leoncavallo AJ, Lukowski ZL, Greer AB, Martorana GM, Zou B, Shuster JJ, Jay Katz L, Schuman JS, Kass MA, Sherwood MB. Comparing glaucomatous disc change using stereo disc viewing and the MatchedFlicker programme in glaucoma experts and trainees. Br J Ophthalmol. 2018 Mar;102(3):358-363. doi: 10.1136/bjophthalmol-2017-310336. Epub 2017 Aug 16. PMID 28814418
- [Background] Gao F, Philip Miller J, Xiong C, Luo J, Beiser JA, Chen L, Gordon MO. Estimating correlation between multivariate longitudinal data in the presence of heterogeneity. BMC Med Res Methodol. 2017 Aug 17;17(1):124. doi: 10.1186/s12874-017-0398-1. PMID 28818061
- [Background] Chen Z, Wang K. A gene-based test of association through an orthogonal decomposition of genotype scores. Hum Genet. 2017 Oct;136(10):1385-1394. doi: 10.1007/s00439-017-1839-y. Epub 2017 Sep 1. PMID 28864915
- [Background] Wang K. Conditional asymptotic inference for the kernel association test. Bioinformatics. 2017 Dec 1;33(23):3733-3739. doi: 10.1093/bioinformatics/btx511. PMID 28961861
- [Background] Gordon MO, Kass MA. What We Have Learned From the Ocular Hypertension Treatment Study. Am J Ophthalmol. 2018 May;189:xxiv-xxvii. doi: 10.1016/j.ajo.2018.02.016. Epub 2018 Mar 1. PMID 29501371
- [Background] Gordon MO, Higginbotham EJ, Heuer DK, Parrish RK 2nd, Robin AL, Morris PA, Dunn DA, Wilson BS, Kass MA; Ocular Hypertension Treatment Study. Assessment of the Impact of an Endpoint Committee in the Ocular Hypertension Treatment Study. Am J Ophthalmol. 2019 Mar;199:193-199. doi: 10.1016/j.ajo.2018.11.006. Epub 2018 Nov 22. PMID 30471242
- [Derived] Sekimitsu S, Ghazal N, Aziz K, Zhao Y, Singh RK, Fingert JH, Gordon MO, Kass MA, Scheetz T, Segre AV, Pasquale LR, Wiggs JL, Brandt JD, Zebardast N. Primary Open-Angle Glaucoma Polygenic Risk Score and Risk of Disease Onset: A Post Hoc Analysis of a Randomized Clinical Trial. JAMA Ophthalmol. 2024 Nov 7;142(12):1132-9. doi: 10.1001/jamaophthalmol.2024.4376. Online ahead of print. PMID 39509108
- [Derived] Singh RK, Zhao Y, Elze T, Fingert J, Gordon M, Kass MA, Luo Y, Pasquale LR, Scheetz T, Segre AV, Wiggs JL, Zebardast N. Polygenic Risk Scores for Glaucoma Onset in the Ocular Hypertension Treatment Study. JAMA Ophthalmol. 2024 Apr 1;142(4):356-363. doi: 10.1001/jamaophthalmol.2024.0151. PMID 38483402
- [Derived] Gao F, Luo J, Liu J, Wan F, Wang G, Gordon M, Xiong C. Comparing statistical methods in assessing the prognostic effect of biomarker variability on time-to-event clinical outcomes. BMC Med Res Methodol. 2022 Jul 22;22(1):201. doi: 10.1186/s12874-022-01686-7. PMID 35869438
- [Derived] Kass MA, Heuer DK, Higginbotham EJ, Parrish RK, Khanna CL, Brandt JD, Soltau JB, Johnson CA, Keltner JL, Huecker JB, Wilson BS, Liu L, Miller JP, Quigley HA, Gordon MO; Ocular Hypertension Study Group. Assessment of Cumulative Incidence and Severity of Primary Open-Angle Glaucoma Among Participants in the Ocular Hypertension Treatment Study After 20 Years of Follow-up. JAMA Ophthalmol. 2021 Apr 15;139(5):1-9. doi: 10.1001/jamaophthalmol.2021.0341. Online ahead of print. PMID 33856434
- [Derived] Kass MA, Gordon MO, Gao F, Heuer DK, Higginbotham EJ, Johnson CA, Keltner JK, Miller JP, Parrish RK, Wilson MR; Ocular Hypertension Treatment Study Group. Delaying treatment of ocular hypertension: the ocular hypertension treatment study. Arch Ophthalmol. 2010 Mar;128(3):276-87. doi: 10.1001/archophthalmol.2010.20. PMID 20212196

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Topical ocular hypotensive eye drops.
Period: Overall Study
Arm/Group | Observation | Treatment
Started | 819 | 817
Completed OHTS Phase I, June 2002 | 706 | 702
Completed | 580 (Completed OHTS Phase 2, through March 2009) | 579 (Completed OHTS Phase 2, through March 2009)
Not Completed | 239 | 238

BASELINE CHARACTERISTICS:
Population: 1636 ocular hypertensive patients were randomized to either close observation or ocular hypertensive medication.
Groups:
- Observation: Observation only
- Treatment: Topical Antiglaucoma Agents: Topical Antiglaucoma Agents
- Total: Total of all reporting groups
Arm/Group | Observation | Treatment | Total
Number analyzed (Participants) | 819 | 817 | 1636
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (9.7) | 55.2 (9.5) | 55.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 346 | 359 | 705
  Male | 473 | 458 | 931
Race/Ethnicity, Customized [Number; unit: participants]
  Native American | 3 | 1 | 4
  Asian | 10 | 4 | 14
  African American | 205 | 203 | 408
  Hispanic | 35 | 24 | 59
  White | 560 | 577 | 1137
  Other | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Primary Open-Angle Glaucoma in Hypotensive Patients
Description: Comparison of the cumulative proportion of participants who develop primary open-angle glaucoma in the observation and medication groups.
Time Frame: 5 yrs (OHTS I, June 2002) and 13.0 yrs (completion of both phases of OHTS, March 2009)
Population: 1636 ocular hypertensive participants were randomized to either close observation or treatment with topical hypotensive eyedrops from February 1994 through June 2002. In June 2002 the observation participants were offered treatment with topical hypotensive eyedrops.
Measure: Number; unit: percent of participants
Groups:
- Observation: Observation only from February 1994 through June 2002.Observation participants were offered topical antiglaucoma agents after June 2002 through study close out March 2009.
- Treatment: Topical ocular hypotensive eye drops from February 1994 through March 2009.
Arm/Group | Observation | Treatment
Number analyzed (Participants) | 819 | 817
percent of participants
  Incidence of glaucoma at 5 yr (OHTS I, June 2002) | 9.5 | 4.4
  Incidence of glaucoma 13 yr (OHTS II, March 2009) | 20.0 | 14.1

ADVERSE EVENTS:
Time Frame: Adverse events collected during OHTS I, from February 1994 to June 2002.
Description: Specific ocular adverse events are unknown because adverse events were only collected with regard to organ system.
Groups:
- Observation: Observation only from February 1994 to June 2002 .
- Treatment: Topical Antiglaucoma Agents: Topical Antiglaucoma Agents from February 1994 to June 2002.
Arm/Group | Observation | Treatment
Serious Adverse Events (participants affected / at risk) | 12/819 | 13/817
Other Adverse Events (participants affected / at risk) | 481/819 | 570/817
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Observation (N=819) | Treatment (N=817)
Ocular Serious Adverse Events (OHTS I, June 2002) (Eye disorders) | 12 | 13 — Specific ocular serious adverse events are unknown because they were only collected with regard to organ system.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Observation (N=819) | Treatment (N=817)
Ocular Adverse Event (Not Serious) (Eye disorders) | 481 | 570 — Adverse Events that were not serious.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Informed Consent Form (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT00000125/ICF_000.pdf